CLINICAL TRIAL: NCT07339631
Title: The Safety and Clinical Efficacy of Sodium Aescinate: A Double-Blind, Randomized Controlled Trial for the Treatment of Low Back Pain (LBP) in Adults
Brief Title: Sodium Aescinate for the Treatment of Low Back Pain (LBP) in Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Bo Gao, MD, principal investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20252323
Record Dates: First submitted 2025-12-22; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain; Paraspinal Muscle; CLBP - Chronic Low Back Pain; Non-specific Chronic Low Back Pain
Keywords: low back pain; sodium aescinate tablets; double-blind randomized controlled trial; CLBP - Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — sodium aescinate

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective parallel-group study. Participants are randomly assigned to either the experimental group (sodium aescinate tablets) or the placebo group in a 1:1 ratio. Both groups receive the assigned intervention for 6 consecutive weeks, with no crossover between groups during the study period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A dedicated researcher (not involved in data collection, analysis, or follow-up) prepares and distributes the study medications (sodium aescinate tablets and matching placebo), which are identical in appearance, dosage form, and administration route to ensure masking. Emergency unblinding is permitted for safety reasons, with documentation of the date and reason required within 48 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in this arm will receive oral sodium aescinate mimetic tablets (placebo), which are identical to the experimental drug (sodium aescinate tablets) in appearance, dosage form, color, and taste.
  Interventions: Drug: Placebo
- Sodium Aescinate Tablets (Experimental): Participants in this arm will receive oral sodium aescinate tablets.
  Interventions: Drug: Sodium Aescinate Tablets

INTERVENTIONS:
Drug: Sodium Aescinate Tablets — This intervention is an oral sodium aescinate tablets. Each tablet contains 30mg of sodium aescinate as the active ingredient. Eligible participants will take 2 tablets per dose, twice daily (bid), for a continuous 6-week treatment period. The drug is provided by Shandong Luye Pharmaceutical Co., Ltd. and is administered in a double-blind manner, with the placebo control having identical appearance, dosage form, and administration route to ensure masking. The intervention aims to improve pain, disability, and functional status in adult patients with chronic low back pain by exerting anti-inflammatory, detumescent, and microcirculation-improving effects.
  Arms: Sodium Aescinate Tablets
Drug: Placebo — The intervention dosage is 2 tablets (30mg/tablet) per administration, twice daily (bid), for a continuous 6-week treatment period. During the study, participants will complete follow-up visits at baseline (week 0), week 1, week 3, and week 6 for efficacy assessments (VAS, ODI, JOA, SF-36 scores) and undergo lumbar MRI scans at baseline and week 6 to measure paraspinal muscle cross-sectional area and fat infiltration rate. All adverse events experienced during the treatment period will be recorded in detail.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the clinical efficacy and safety of sodium aescinate in treating low back pain (LBP) in adult participants.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of oral sodium aescinate in improving symptoms and function in adult participants aged 18-65 years with low back pain (LBP) lasting at least 12 weeks and a Visual Analog Scale (VAS) score > 4 points. The main questions it aims to answer are:

1. Does oral sodium aescinate tablets reduce pain intensity (measured by VAS score) in adult LBP patients at 1, 3, and 6 weeks after treatment?
2. Is oral sodium aescinate tablets safe for adult LBP patients, with an acceptable adverse event profile during the 6-week treatment period?

Researchers will compare participants receiving sodium aescinate (experimental group) to those receiving a placebo (control group) to see if the experimental intervention results in significant improvements in pain, disability, functional status, and lumbar paraspinal muscle conditions (cross-sectional area and fat infiltration rate) compared to the placebo.

Participants will:

1. Undergo screening (medical history review, physical examination, and relevant tests) to confirm eligibility and sign an informed consent form.
2. Be randomly assigned to either the experimental or control group in a 1:1 ratio.
3. Take 2 tablets of the assigned study medication (sodium aescinate tablets or placebo) twice daily for 6 consecutive weeks.
4. Complete follow-up visits at baseline (week 0), week 1, week 3, and week 6 for efficacy assessments (VAS, Oswestry Disability Index [ODI], Japanese Orthopaedic Association [JOA] score, 36-Item Short Form Health Survey [SF-36] score).
5. Undergo lumbar MRI scans at baseline and week 6 to measure paraspinal muscle cross-sectional area and fat infiltration rate.
6. Report any adverse events experienced during the 6-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for chronic low back pain (cLBP) recommended by the Clinical Practice Guidelines for Chronic Low Back Pain in China (2024 Edition): the course of disease lasts at least 12 weeks, with pain occurring in the region below the lower costal margin, above the gluteal crease (horizontal gluteal fold), and between the midaxillary lines on both sides, which may be accompanied by pain in one or both lower extremities.
2. Has moderate to severe pain, with a Visual Analog Scale (VAS) score > 4 points.
3. Aged between 18 and 65 years old.
4. Has a clear understanding of the study content, good compliance, and high willingness to cooperate.
5. Has signed a written informed consent form voluntarily.

Exclusion Criteria:

1. Is in the acute pain phase or acute exacerbation of chronic pain.
2. Has low back pain caused by other reasons such as infectious diseases or tumors, including but not limited to spinal tumors, spinal tuberculosis, spinal cord infections, etc.
3. Has a history of allergy to sodium aescinate.
4. Suffers from systemic diseases or organ dysfunction.
5. Has participated in other clinical trials within 1 month before enrollment.
6. Has severe mental illness or other conditions that prevent cooperation with the study.
7. Is a pregnant or lactating woman, or a woman planning to become pregnant.
8. Has metal implants or other conditions that are not suitable for MRI examination.
9. Is considered by the researcher to have conditions that are unfavorable for completing the study course.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Assessed by Visual Analog Scale (VAS) Score | Baseline (Day 0, pre-intervention), Week 1, Week 3, and Week 6 after the start of treatment
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated tool with a score range from 0 to 10 points. A score of 0 represents no pain, and a score of 10 represents the most severe pain imaginable. This outcome measure evaluates changes in pain intensity in adults with chronic low back pain (cLBP) following treatment with oral sodium aescinate tablets.

SECONDARY OUTCOMES:
Disability Severity Assessed by Oswestry Disability Index (ODI) Score | Baseline (Day 0, pre-intervention), Week 1, Week 3, and Week 6 after the start of treatment
  Disability related to low back pain will be assessed using the Oswestry Disability Index (ODI), a widely used questionnaire with a total score range of 0 to 50 points. Higher scores indicate greater disability in activities of daily living. This outcome measure evaluates changes in functional disability in cLBP patients after treatment.
Lumbar Functional Status Assessed by Japanese Orthopaedic Association (JOA) Score | Baseline (Day 0, pre-intervention), Week 1, Week 3, and Week 6 after the start of treatment
  Lumbar spine function will be evaluated using the Japanese Orthopaedic Association (JOA) score, which ranges from 0 to 29 points. Lower scores indicate more severe functional impairment. This outcome measure assesses changes in lumbar spine function following treatment.
Health-Related Quality of Life Assessed by SF-36 Total Score | Baseline (Day 0, pre-intervention), Week 1, Week 3, and Week 6 after the start of treatment
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). The total score ranges from 0 to 100 points, with higher scores indicating better overall health status. This outcome measure evaluates changes in overall quality of life in cLBP patients following treatment.
Lumbar Paraspinal Muscle Cross-Sectional Area Assessed by MRI | Baseline (Day 0, pre-intervention) and Week 6 after the start of treatment
  Lumbar MRI will be used to measure the cross-sectional area of paraspinal muscles as an objective indicator of muscle mass. This outcome measure evaluates changes in paraspinal muscle size following treatment with sodium aescinate tablets.
Lumbar Paraspinal Muscle Fat Infiltration Rate Assessed by MRI | Baseline (Day 0, pre-intervention) and Week 6 after the start of treatment
  Lumbar MRI will be used to assess the fat infiltration rate of paraspinal muscles as an indicator of muscle quality. This outcome measure evaluates changes in paraspinal muscle composition following treatment.

OTHER OUTCOMES:
Incidence of Adverse Events During Treatment | Within 6 weeks after the start of treatment
  All adverse events (AEs) occurring during the 6-week treatment period will be recorded. For each AE, the type, severity, duration, and relationship to the study drug will be documented to evaluate the safety of oral sodium aescinate tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Xjing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No